CLINICAL TRIAL: NCT02645136
Title: The Effects of Pilates Method in Muscle Strength of the Pelvic Floor as Treatment of Post Prostatectomy Urinary Incontinence: : a Randomized Control Trial
Brief Title: The Effects of Pilates in Muscle Strength of the Pelvic Floor as Treatment of Post Prostatectomy Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Cíntia Spagnolo Gomes, Physioterapist student of a masters degree program at the Center of Health Science, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 820.529
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PILATES (Experimental): Weekly Pilates sessions, guided by a specialized physiotherapist. The duration of the treatment was 10 weeks, and each session lasted 45 to 50 minutes. All subjects received instruction to perform specific daily home exercises.
  Interventions: Other: Pilates
- PFMT and AES (Active Comparator): For also 10 weeks, the participants went trough anal electrical stimulation (AES) associated with Pelvic Floor Muscle Training (PFMT), supervised by a specialized physiotherapist. All subjects received orientation to perform the same pelvic floor exercises at home.
  Interventions: Other: PFMT and AES
- Control (Placebo Comparator): Control Group
  Interventions: Other: Control

INTERVENTIONS:
Other: Pilates — Pilates exercises
  Arms: PILATES
Other: PFMT and AES — conventional pelvic floor muscle exercises combined with anal electrical stimulation Device: electrical stimulation (Dualpex 961 Uro®)
  Arms: PFMT and AES
Other: Control
  Arms: Control

SUMMARY:
The purpose of this study is to compare the efficacy between a Pilates exercise program and a Pelvic Floor Muscle Training (PFMT) protocol combined with anal electrical stimulation (AES) in muscular pressure strength of the pelvic floor as conservative treatment of urinary incontinence after prostatectomy.

DETAILED DESCRIPTION:
This randomized clinical trial includes 115 individuals with urinary incontinence one month after radical prostatectomy. One physiotherapist, with experience in urogynecology, was responsible for all the assessments. muscular pressure strength of the pelvic floor, 24-hour pad test and the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) were the variables evaluated.

The subjects were allocated in one of three treatment groups (G1: Pilates; G2: anal electrical stimulation combined with pelvic floor muscle training and G3: Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 50 and 75 years old;
* Submitted to radical prostatectomy;
* With complaints of urinary incontinence;
* That completed one month of surgery;

Exclusion Criteria:

* History of incontinence;
* Transurethral resection of the prostate;
* Diagnosis of neurological or cognitive impairment;
* Subjects who were unable to attend treatment sessions, due to distance or physical limitations.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
improves muscle strength of the pelvic floor at 3 months | baseline and 3 months
  Evaluation of the contraction capacity of the pelvic floor using perineometer (Myomed 932 Enraf/Nonius®)

SECONDARY OUTCOMES:
Change in the International Consultation of Urinary Incontinence- Short Form questionnaire at 3 months | baseline and 3 months
Change in Pad test 24 hours at 3 months | baseline and 3 months

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660
- [Derived] Gomes CS, Pedriali FR, Urbano MR, Moreira EH, Averbeck MA, Almeida SHM. The effects of Pilates method on pelvic floor muscle strength in patients with post-prostatectomy urinary incontinence: A randomized clinical trial. Neurourol Urodyn. 2018 Jan;37(1):346-353. doi: 10.1002/nau.23300. Epub 2017 May 2. PMID 28464434